CLINICAL TRIAL: NCT01202526
Title: The Effect of Roux-en-Y Gastric Bypass on Insulin Sensitivity in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anna Kirstine Bojsen-Moeller, MD, Hvidovre University Hospital
Other Study IDs: ISBypass
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Insulin resistance; Gastric bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine, muscle, subcutaneous fat, visceral fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RYGB patients with type 2 diabetes: Morbid obese patients with type 2 diabetes undergoing gastric bypass surgery
- RYGB patients without type 2 diabetes: Morbid obese patients with normal glucose tolerance undergoing gastric bypass surgery

SUMMARY:
Gastric bypass surgery induces remission of diabetes within days after surgery, before significant weight loss. The aim of the study is to examine whether improved insulin sensitivity of muscle and liver contributes to the immediate diabetes resolution.

DETAILED DESCRIPTION:
Obesity has become a severe epidemic globally. With the rapid increase in obesity comes a pronounced rise in obesity-related disorders, especially type 2 diabetes. Weight loss achieved through lifestyle changes improves diabetes, but is very difficult to maintain over time. In contrast, Roux-en-Y gastric bypass (RYGB) surgery can induce long-term weight loss and remission of diabetes. Surprisingly, the resolution of type 2 diabetes occurs within days after surgery and before significant weight loss. The resolution of diabetes must therefore be explained by a response to the surgical alterations of the stomach and intestines: restriction in gastric volume and bypass of the stomach, duodenum and proximal jejunum.

Severe insulin resistance in muscle and liver is the common defect in obesity and type 2 diabetes and may be improved or even reversed shortly after the operation. The aim of this study is to examine the acute changes in insulin sensitivity of muscle and liver by using hyperinsulinaemic euglycaemic clamp combined with glucose tracer to assess hepatic glucose production. Insulin signaling pathways will be studied in biopsies from muscle and subcutaneous fat as to explain the molecular basis of the changes in insulin sensitivity after RYGB.

Insulin secretion will be evaluated in response to oral glucose as well as iv glucose-glucagon.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for gastric bypass surgery
* Verified type 2 diabetes or normal glucose tolerance by oral glucose tolerance test (OGTT)

Exclusion Criteria:

* Treatment for Hyperthyroidism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are recruited from the outpatient clinic of endocrinology and gastrosurgical clinic at Hvidovre University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity after RYGB | 1 week, 3 months, 1 year

SECONDARY OUTCOMES:
Change in insulin secretion in response to oral glucose after RYGB | 3 months, 1 year

OTHER OUTCOMES:
Change in insulin secretion after iv glucose-glucagon after RYGB | 1 week, 3months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kirstine Bojsen-Møller, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Wewer Albrechtsen NJ, Hartmann B, Veedfald S, Windelov JA, Plamboeck A, Bojsen-Moller KN, Idorn T, Feldt-Rasmussen B, Knop FK, Vilsboll T, Madsbad S, Deacon CF, Holst JJ. Hyperglucagonaemia analysed by glucagon sandwich ELISA: nonspecific interference or truly elevated levels? Diabetologia. 2014 Sep;57(9):1919-26. doi: 10.1007/s00125-014-3283-z. Epub 2014 Jun 3. PMID 24891019
- [Derived] Bojsen-Moller KN, Dirksen C, Jorgensen NB, Jacobsen SH, Serup AK, Albers PH, Hansen DL, Worm D, Naver L, Kristiansen VB, Wojtaszewski JF, Kiens B, Holst JJ, Richter EA, Madsbad S. Early enhancements of hepatic and later of peripheral insulin sensitivity combined with increased postprandial insulin secretion contribute to improved glycemic control after Roux-en-Y gastric bypass. Diabetes. 2014 May;63(5):1725-37. doi: 10.2337/db13-1307. Epub 2013 Nov 15. PMID 24241533